CLINICAL TRIAL: NCT01074957
Title: Effects of Physical Therapy on Pulmonary Volumes
Brief Title: Effects of Physical Therapy on Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Universitário Augusto Motta (Other)
Responsible Party: Cristina Márcia Dias, Centro Universitário Augusto Motta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UNISUAM; Mestrado UNISUAM (Other: UNISUAM)
Record Dates: First submitted 2010-02-22; First posted 2010-02-24 (Estimated); Last update posted 2010-02-24 (Estimated); Status verified 2010-02

CONDITIONS: Pulmonary Volumes After Cardiac Surgery
MeSH Terms: interventions — Exercise; Early Ambulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Incentive Spirometry (Active Comparator): Incentive Spirometry group (IS) was oriented to take a deep breathing through Voldyne 5000TM (Sherwood Medical; St Loius, MO, USA) from Functional Residual Capacity (FRC) to Total Lung Capacity (TLC).
  Interventions: Device: Incentive Spirometry
- Exercise group (Active Comparator): Patients were taught huffing (forced expiration while the glottis is opened), supported cough (with patient's hands placed on the sternotomy incision) and mobilization, including active limb exercises, sit out of bed and deambulation (starting on the third postoperative day).
  Interventions: Other: Exercise
- Breath-Stacking (Active Comparator): Breath-Stacking group (BS) performed successive inspiratory efforts using a facial mask adapted to an unidirectional valve
  Interventions: Device: Breath-Stacking Technique

INTERVENTIONS:
Device: Incentive Spirometry — Incentive Spirometry (IS) has been used extensively in postoperative period and consists of spontaneous deep breaths through a device which provides a visual feedback to maintain a maximum insuflation
  Other Names: Voldyne
  Arms: Incentive Spirometry
Device: Breath-Stacking Technique — An one-way valve device to promote the summation of successive inspiratory volumes while expiration was avoided
  Other Names: One-way inspiratory valve
  Arms: Breath-Stacking
Other: Exercise — Patients were taught huffing (forced expiration while the glottis is opened), supported cough (with patient's hands placed on the sternotomy incision) and mobilization, including active limb exercises, sit out of bed and deambulation (starting on the third postoperative day).
  Other Names: Early mobilization
  Arms: Exercise group

SUMMARY:
Background: Although respiratory physiotherapy has been used in patients undergoing cardiac surgery, evidence lacks concerning its effectiveness. The aim of this study was to evaluate the efficacy of three physiotherapeutic protocols used to recover respiratory volumes in the postoperative period.

Methods: Thirty five patients were randomly allocated into three groups. Exercise group (E) was oriented to progressive mobilization. Incentive Spirometry group (IS) performed deep breathings using VoldyneTM, while Breath-Stacking group (BS) performed successive inspiratory efforts using a facial mask adapted to an unidirectional valve. Both BS and IS also performed progressive mobilization. Forced spirometry was carried out in the pre-operative period and from the first to the fifth postoperative day. Statistical analysis used student t-test and ANOVA, and the differences were considered significant when p<0.05.

DETAILED DESCRIPTION:
This was a prospective, controlled and randomized clinical trial, conducted with patients undergoing cardiac surgery at Hospital de Força Aérea do Galeão (HFAG - Rio de Janeiro, RJ, Brazil). According to Helsinki declaration, the protocol was approved by UNISUAM Ethics Committee (process: 15/2007) and written informed consent was obtained from all participants. All patients at the HFAG, who were scheduled for cardiac surgery between November 2007 and February 2009 were eligible to participate in this study.

Patients were not included if any of the following criteria was present: informed consent could not be obtained, they could not perform the preoperative tests, cognitive impairments to perform the IS, intolerance to the use of BS mask. Exclusion criteria included: hemodynamic complications (intraoperative myocardial infarction, major blood loss, marked hypotension, reduced cardiac output requiring the use of an intra-aortic balloon pump or extraordinary use of medications) and intubation period longer than 72 hours following arrival in the intensive care unit. In all patients the surgical procedure was through a median sternotomy, and the postoperative routine was the same, including optimal treatment for pain control. A verbal pain score was obtained using a visual analog scale and all patients initiated the physiotherapeutic treatment at the first postoperative day, following extubation. Demographic data, clinical history and preoperative risk factors were recorded.

In the preoperative period all patients were instructed about the importance of early mobilization and excessive bronchial secretion removal. Patients were taught huffing (forced expiration while the glottis is opened), supported cough (with patient's hands placed on the sternotomy incision) and mobilization, including active limb exercises, sit out of bed and deambulation (starting on the third postoperative day). Then, they were randomly allocated into three groups. Exercise group (E) performed only the procedures described above. Incentive Spirometry group (IS) was oriented to take a deep breathing through Voldyne 5000TM (Sherwood Medical; St Loius, MO, USA) from Functional Residual Capacity (FRC) to Total Lung Capacity (TLC). Breath-Stacking group (BS) performed inspiratory efforts using a facial mask adapted to an unidirectional valve. Since the mask was set to allow only inspiration (the expiratory branch was occluded), the patient carried through successive inspiratory efforts for a period of 20 seconds. Then, the expiratory branch was released allowing exhalation. These three treatments were applied for five days, with three series of five maneuvers twice a day. Patients management was similar among groups in terms of assessment, mobilization protocol and cough orientation.

For safety purposes, vital signs and oxygen saturation (SpO2) were monitored throughout the interventions. SpO2 was measured continuously for seven minutes using a portable pulse oximeter (Model 2500A, Nonin Medical INC; Plymouth, USA) with patient breathing room air. After seven minutes the most consistent value for 30 seconds was recorded and previous oxygen therapy was reinitiated. If during the assessment, patient's SpO2 dropped to below 85%, oxygen was recommenced and it was registered.

All procedures were performed under the supervision of an experienced physical therapist. Forced spirometry was carried out in the preoperative period and from the first to the fifth postoperative day, using a Pony Fx® spirometer (Cosmed; Rome, Italy). A Wright® ventilometer (British Oxygen Company; London, England) was properly attached to Voldyne and to Breath-Stacking mask, allowing to measure the Inspiratory Capacity (IC) during the procedures.

Postoperative risk was evaluated by means of Torrington Scale, using clinical and functional data.

Statistical Analysis Statistical analysis was done using Sigma Stat 3.1 (Jandel Scientific, San Rafael, CA, USA). Data are presented as average and standard error of the mean. They presented normal distributions (Kolmogorov-Smirnov test with Lilliefors' correction) and homogeneous variances (Levene median test). Comparisons of FVC between IS, BS and E were done with ANOVA, followed by Tukey test whenever multiple comparisons were required. Student's t-test was used to compare IC between IS and BS. The significance level was always set at 5%.

ELIGIBILITY:
Inclusion Criteria:

Patients were not included if any of the following criteria was present:

* Informed consent could not be obtained
* Could not perform the preoperative tests
* Cognitive impairments to perform the IS
* Intolerance to the use of BS mask

Exclusion Criteria:

Exclusion criteria included:

* Hemodynamic complications (intraoperative myocardial infarction
* Major blood loss
* Marked hypotension
* Reduced cardiac output requiring the use of an intra-aortic balloon pump or extraordinary use of medications) and intubation period longer than 72 hours following arrival in the intensive care unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-11; Primary Completion 2009-07 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Respiratory volume | First five postoperative days

CONTACTS AND LOCATIONS:
Overall Officials: Cristina M Dias, DSc, Principal Investigator — Centro Universitário Augusto Motta